CLINICAL TRIAL: NCT06940466
Title: A Cognitive Intervention to Manage 'Brain Fog' in Menopause Transition: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167427
Record Dates: First submitted 2025-04-03; First posted 2025-04-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Menopause

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treatment group participants will complete a 4 x 2-hour intervention. Key components will include education about menopause and cognition, cognitive strategies (memory, attention and executive functioning), CBT techniques and emotional support
  Interventions: Other: Online cognitive intervention
- Control group (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Online cognitive intervention — A 4 x 2-hour intervention with the following key components: education about menopause and cognition, cognitive strategies (memory, attention and executive functioning), CBT techniques and emotional support.
  Arms: Treatment group

SUMMARY:
Cognitive complaints at menopause transition (MT), often described as 'brain fog'; can include difficulty recalling words and numbers, misplacing items, trouble concentrating and forgetfulness. Whilst these difficulties resolve for most people, several years of reduced cognitive functioning can be highly damaging and result in problems including leaving work, depression and relationship breakdown.

Study Aims: This project aims 1) to develop and finalise a cognitive intervention for the menopause, 2) To evaluate the feasibility, acceptability and preliminary effects of the intervention. 3) To evaluate the interventions preliminary effects on subjective and objective cognition

Relevance: Traditionally Menopause Hormone Therapy (MHT) is offered to women with cognitive complaints due to its beneficial effect. However, many women are unable to take it due to medical reasons or choose not to. If this intervention is concluded as feasible and acceptable it may then be appropriate to conduct a full RCT of this intervention. It could reduce excess disability, potentially enabling people to remain at work and function better in daily life. Costs to the NHS might be reduced through decreased service and medication use.

ELIGIBILITY:
Inclusion Criteria:

* people with ovaries (women, trans-men and non-binary people) aged 40-60
* late-reproductive, early-late perimenopause or early post-menopause stages according to the Stages of Reproductive Aging Workshop (STRAW+10; Harlow et al., 2012)
* stable dose of hormonal (oestrogen, progesterone, testosterone) or antidepressant (SSRI, SSNI) medication for 6 months or more
* self-reported cognitive difficulties impacting on quality of life
* ability to communicate in English

Exclusion Criteria:

* diagnosis of dementia
* new regimen (under 6 months) of medication likely to impact on cognition (i.e. hormonal or anti-depressant)

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Pre-intervention and within 6 weeks post intervention
  The PHQ9 is a self-administered questionnaire measuring levels of depression over the past 2 weeks. The questionnaire uses a 4-point Likert rating scale, ranging from 0 (not at all) to 3 (nearly every day). The total score can range from 0 to 27, with high scores meaning high depression.
Generalised Anxiety Disorder (GAD-7) | Pre-intervention and within 6 weeks post intervention
  The GAD 7 is a self-administered questionnaire measuring levels of anxiety over the past 2 weeks. The questionnaire uses a 4 Likert rating scale, ranging from 0 (not at all) to 3 (nearly every day). Total score can range from 0 to 21 and is categorised by 0-4 was no anxiety, 5-9 was mild anxiety, 10-14 was moderate anxiety, and 15 or above was severe anxiety.
Menopause-Specific Quality of Life (MENQoL) | Pre-intervention and within 6 weeks post intervention
  The MENQoL measures the quality of life over 4 domains of menopausal symptoms: Vasomotor, Psychosocial, Physical and Sexual, asking if a symptom is present or not and if it is to score how bothersome it is on a 7-point Likert scale, ranging from 0 'not bothered at all' to 6 'extremely bothered.
Hot Flush Rating Scale (HFRS) | Pre-intervention and within 6 weeks post intervention
  The HFRS is a self-report measure of the frequency and problem rating of hot flashes and night sweats (also known as vasomotor symptoms [VMS]) over the past week.
The Multifactoral Memory Questionnaire (MMQ) | Pre-intervention and within 6 weeks post intervention
  The MMQ measures self-reported cognitive functions with three subscales: abilities, contentment, strategies. Items are rated on a 5-point scale (0-4), lower scores indicate worse perceived memory.
Menopause-specific Cognitive Scale (MENO-Cog) | Pre-intervention and within 6 weeks post intervention
  The measure is in development with a PhD student in the same research team. It measures self-reported cognition functioning with a 5-point Likert scale; higher scores indicate worse perceived cognitive function.
Rey Auditory Verbal Learning Test (RAVLT) | Pre-intervention and within 6 weeks post intervention
  The RAVLT is a neuropsychological test measuring verbal learning and (immediate and delayed) verbal memory.
Trail Making Test (TMT) | Pre-intervention and within 6 weeks post intervention
  The TMT (Part A and B) is a neuropsychological test assessing executive function; shorter reaction times indicate better performance.
Digit Span subtest (WISC-V) | Pre-intervention and within 6 weeks post intervention
  The Digit Span test (backward and forward) is a neuropsychological test assessing attention and working memory.
Controlled Word Association Test | Pre-intervention and within 6 weeks post intervention
  The Controlled Word Association Test is a neuropsychological test assessing verbal fluency.

SECONDARY OUTCOMES:
Post intervention interviews | Pre-intervention and within 6 weeks post intervention
  Around 15 participants will be invited to qualitative semi-structured audio-recorded interviews to explore their feedback of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No